CLINICAL TRIAL: NCT03567317
Title: Mechanisms of Weight Gain During CPAP Treatment in Patients With Obstructive Sleep Apnea
Brief Title: Weight Gain After CPAP Treatment in Patients With Obstructive Sleep Apnea
Acronym: OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Pedro Rodrigues Genta, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: weightgain
Record Dates: First submitted 2018-06-11; First posted 2018-06-25 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: CPAP; Weight Gain; obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP (No Intervention): According to study design, patients will be randomized to remain on CPAP during the initial study visit or withdraw CPAP one week before. If randomized to withdraw CPAP during the initial study visit, patients will resume CPAP use for one week before the second study visit.
- CPAP withdrawal (Experimental): According to study design, patients will be randomized to remain on CPAP during the initial study visit or withdraw CPAP one week before. If randomized to withdraw CPAP at the second study visit, patients will withdraw CPAP one week before.
  Interventions: Device: CPAP withdrawal

INTERVENTIONS:
Device: CPAP withdrawal — Patients randomized to withdrawal will stop CPAP use for one week before study evaluations. Patients will also undergo a polysomnography to confirm the presence of severe OSA.
  Arms: CPAP withdrawal

SUMMARY:
The purpose of this trial is to investigate the mechanisms leading to weight gain during CPAP treatment for obstructive sleep apnea (OSA).

DETAILED DESCRIPTION:
Obesity and obstructive sleep apnea share a bidirectional relationship. While obesity is a major risk factor for OSA, OSA may contribute to weight gain. Recent evidence suggests that OSA treatment is associated with weight gain. The mechanisms involved in weight gain after OSA treatment are not known. The purpose of this study is to determine the mechanisms of weight gain during CPAP treatment for severe OSA leads. The investigators hypothesis is that CPAP leads to a decrease in energy expenditure and prevents the elimination of extracellular fluid that is accumulated during the day. In order to test this hypothesis, 20 patients with severe OSA aged between 50 and 80 years old, under regular treatment with CPAP, will be invited to participate. Using a cross-over design, the investigators will perform bioelectric impedance 5 times over 24 hours in order to assess the circadian effect of fluid accumulation in two different conditions: during CPAP treatment and 7 days after CPAP withdrawal. A full polysomnography will be performed during CPAP withdrawal to confirm severe OSA and during CPAP treatment to confirm adequate control of respiratory events. In addition, basal metabolic rate, hematocrit, serum BNP, urinary sodium, creatinine and osmolality will be determined in the morning during the CPAP and CPAP withdrawal periods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of severe OSA (AHI>30 events/h)
* 50 and 80 years old
* regular treatment with CPAP with an average daily use of >4hours

Exclusion Criteria:

* congestive heart failure
* renal insufficiency
* hepatic failure
* urinary incontinency
* diuretic therapy

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Extracellular fluid volume | Seven days
  Extracellular fluid volume accumulation will be assessed by bioelectrical impedance after 7 days of CPAP or CPAP withdrawal.

SECONDARY OUTCOMES:
Basal metabolic rate | 24 hours
  Basal metabolic rate will be assessed by indirect calorimetry after 7 days of CPAP or CPAP withdrawal.
Weight change | 7 days
  Weight change during CPAP use

CONTACTS AND LOCATIONS:
Overall Officials: Pedro R Genta, MD, Principal Investigator — Sleep Laboratoy, Heart Institute
Locations (1):
- Sleep Laboratory, Heart Institute, Pulmonary Division, Hospital das Clínicas da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Herculano S, Grad GF, Drager LF, de Albuquerque ALP, Melo CM, Lorenzi-Filho G, Genta PR. Weight Gain Induced by Continuous Positive Airway Pressure in Patients with Obstructive Sleep Apnea Is Mediated by Fluid Accumulation: A Randomized Crossover Controlled Trial. Am J Respir Crit Care Med. 2021 Jan 1;203(1):134-136. doi: 10.1164/rccm.202005-1853LE. No abstract available. PMID 32857590